CLINICAL TRIAL: NCT07003789
Title: Co-Developing a Women-Centered HIV Prevention Intervention to Reduce Stigma, Increase HIV Self-Testing, and Improve PrEP Awareness and Uptake in Ghana
Brief Title: Co-Developing an HIV Prevention Program for Women in Ghana
Acronym: WISEWOMAN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Gloria Aidoo-Frimpong, Principal Investigator, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00009328
Record Dates: First submitted 2025-05-12; First posted 2025-06-04 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: HIV Prevention; Women's Health; Sexual and Reproductive Health
Keywords: HIV self-testing (HIVST); Pre-exposure prophylaxis (PrEP); Youth-centered design; Sub-Saharan Africa; AGYW (Adolescent Girls and Young Women); HIV Stigma; Ghana
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Intervention Model Description: A mixed-methods, community-based participatory intervention. Participants co-develop the HIV prevention program and then pilot test it through WhatsApp-based activities.
Masking Description: No masking is used in this study. All participants and study staff are aware of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women-Centered HIV Prevention Group (Experimental): Participants will take part in a co-developed HIV prevention intervention created through participatory workshops. The intervention will be delivered via WhatsApp over 4 weeks and will include HIV prevention messaging, discussion prompts, and peer support to improve awareness and uptake of HIV self-testing (HIVST) and pre-exposure prophylaxis (PrEP), and reduce stigma.
  Interventions: Behavioral: Women-Centered HIV Prevention Program

INTERVENTIONS:
Behavioral: Women-Centered HIV Prevention Program — This behavioral intervention consists of a participatory, youth-designed HIV prevention program that uses Human-Centered Design (HCD) principles and WhatsApp-based engagement. It includes information and support for HIV self-testing and PrEP, with the goal of increasing awareness, improving uptake, and reducing stigma among young women in Ghana.

SUMMARY:
The WISE Woman Study is a research project in Ghana focused on improving HIV prevention among young women aged 18 to 35. In Ghana, young women are at higher risk of HIV but often lack access to the right information and services. This study will first work with young women and community partners to co-develop a youth-friendly and women-centered HIV prevention program. The program will focus on two proven strategies: HIV self-testing (HIVST) and pre-exposure prophylaxis (PrEP), a medicine that helps prevent HIV.

After the program is created, researchers will test it with 50 young women in Greater Accra and the Eastern Region to see if it's acceptable, easy to use, and if it helps increase knowledge and use of HIVST and PrEP. The intervention will be delivered through WhatsApp and community-based workshops to ensure privacy and reach. Participants will complete surveys and take part in discussions and interviews to share their feedback. This research will help build better HIV prevention strategies tailored to the needs of young women in Ghana.

DETAILED DESCRIPTION:
Young women in Ghana face some of the highest risks of HIV infection in the country, yet they often lack access to HIV prevention tools and supportive services that are tailored to their needs. Many of the barriers they face-including stigma, low awareness, and limited youth-friendly options-can prevent them from accessing HIV self-testing (HIVST) or pre-exposure prophylaxis (PrEP), which are proven prevention methods.

The WISE Woman Study seeks to address these barriers by engaging young women as equal partners in the design and implementation of an HIV prevention intervention. The study is based on the idea that solutions are more effective when they are created with the community, not for it. It uses participatory methods to involve young women in shaping the intervention and includes two main phases:

Phase 1 - Co-Development Workshop:

Fifteen participants-including ten young women and five community stakeholders (such as healthcare workers or peer educators)-will take part in a full-day participatory workshop. During this workshop, they will identify key barriers to HIV prevention, co-create solutions, and help design the structure of the intervention. Structured methods such as the Nominal Group Technique (NGT) and Human-Centered Design (HCD) will be used to ensure that all voices are heard and that the final program reflects the participants' preferences and lived experiences.

Phase 2 - Pilot Study:

Fifty young women aged 18-35 will participate in a 4-week pilot study to test the feasibility and acceptability of the co-developed intervention. Participants will receive information, support, and discussion prompts through WhatsApp-a platform commonly used in Ghana. They will complete short surveys before and after the intervention, and a subset will take part in in-depth interviews to reflect on their experiences. The study will look at changes in knowledge and attitudes toward HIV prevention, willingness to use HIVST and PrEP, and whether participants feel more empowered to take charge of their sexual health.

This study is designed with privacy, respect, and participant safety in mind. By using a mobile platform and focusing on community co-creation, the WISE Woman Study offers an innovative approach to strengthening HIV prevention among young women in Ghana. The findings will help inform future HIV programs and may serve as a model for youth-centered public health interventions in similar settings.

ELIGIBILITY:
Inclusion Criteria:

Identify as female and be between 18-35 years of age

Reside in Greater Accra or the Eastern Region of Ghana

Be sexually active (defined as having engaged in vaginal, anal, or oral sex in the past 6 months)

Have access to a mobile phone with WhatsApp

Be willing to provide informed consent

Be interested in participating in HIV prevention activities

Be comfortable discussing sexual and reproductive health in a group setting (for the workshop)

For pilot phase only: must not have participated in the co-development workshop

Exclusion Criteria:

Do not reside in the two specified regions of Ghana

Unable to provide informed consent

Have cognitive impairments or severe mental health conditions limiting participation

Community partners with commercial conflicts of interest (for workshop only)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility as Measured by FIM Score | Week 5 (end of intervention)
  Feasibility of the intervention will be measured using the Feasibility of Intervention Measure (FIM), a validated 4-item scale. Each item is rated on a 5-point Likert scale (1 = completely disagree to 5 = completely agree). Scores will be summarized using means and standard deviations. Higher scores indicate greater feasibility.
  Unit of Measure: Mean FIM score (1-5 scale)
Acceptability as Measured by AIM Score | Week 5 (post-intervention)
  Acceptability of the intervention will be measured using the Acceptability of Intervention Measure (AIM), a validated 4-item scale with 5-point Likert responses. Scores range from 1 (completely disagree) to 5 (completely agree). Higher scores indicate greater acceptability. Results will be reported as mean and standard deviation.
  Unit of Measure: Mean AIM score (1-5 scale)
Uptake of HIV self-testing (HIVST) | Baseline to Week 8
  Defined as the number of participants who report completing an HIV self-test during the study period, verified via WhatsApp photo confirmation or verbal report.
  Unit of Measure: Number of participants (count)
Willingness to Use PrEP (Survey-Based Behavioral Intention) | Baseline to Week 8
  Willingness will be measured using a validated PrEP intention scale in pre- and post-surveys (e.g., "I am likely to take PrEP in the next 3 months"). Items are scored on a 1 to 5 Likert scale, with higher scores indicating greater willingness to use PrEP. Change in mean intention scores will be reported.
  Unit of Measure: Mean change in score (1-5 scale)
Intervention Completion Rate | Week 5
  Defined as the percentage of participants who complete all required activities during the 4-week WhatsApp-based intervention, including pre- and post-surveys.
  Unit of Measure: Percentage of participants (%)

SECONDARY OUTCOMES:
Reduction in HIV-Related Stigma (Survey Score Change) | Baseline to Week 8
  HIV-related stigma will be measured using an adapted multi-item stigma scale (e.g., internalized and anticipated stigma). Change from pre- to post-intervention will be reported. Scores will be reported as mean change from pre- to post-intervention. The scale ranges from 1 (low stigma) to 5 (high stigma). Lower scores indicate a reduction in stigma (better outcome).
  Unit of Measure: Mean change in stigma score
Number of Participants Reporting the WhatsApp-Based Intervention is Sustainable and Scalable | Week 6-8 (exit interviews)
  Assessed qualitatively via thematic analysis of exit interviews. Participants will be asked if the WhatsApp format and intervention content could be maintained and scaled in their community. Themes will be summarized narratively.
  Unit of Measure: Not applicable - qualitative outcome
Perceived Appropriateness of the Intervention (IAM Score) | Week 5
  Appropriateness of the intervention will be measured using the Intervention Appropriateness Measure (IAM), a validated 4-item scale with 5-point Likert responses. Scores range from 1 (completely disagree) to 5 (completely agree). Higher scores indicate greater perceived appropriateness. Results will be reported as mean and standard deviation.
  Unit of Measure: Mean IAM score (1-5 scale)

CONTACTS AND LOCATIONS:
Overall Officials: Gloria A Aidoo-Frimpong, PhD, MPH, MA, Principal Investigator — SUNY BUFFALO
Locations (1):
- EARC, Accra, Ghana

IPD SHARING:
Plan to Share IPD: No
Due to the sensitive nature of the data related to HIV status, stigma, and participant privacy-especially within a small, community-based sample-individual participant data (IPD) will not be shared to protect confidentiality.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/89/NCT07003789/Prot_SAP_000.pdf